CLINICAL TRIAL: NCT00151593
Title: Celsior®: Evaluation of an Organ Preservation Solution in Liver Transplantation.
Brief Title: Evaluation of Celsior® in Liver Transplant Preservation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Sangstat Medical Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFSSAPS 020007; LOC-H/01-04; CIC0203/006
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Liver Transplantation
Keywords: Cold storage; Liver transplantation; Preservation solution
MeSH Terms: interventions — Celsior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Celsior preservation solution
  Interventions: Other: Celsior®

INTERVENTIONS:
Other: Celsior® — Graft preservation solution

SUMMARY:
The aim of the study is to determine the efficacy and safety of a preservation solution in liver transplantation. Its efficacy will be compared to the efficacy of other currently used preservation solutions.

DETAILED DESCRIPTION:
The quality of organ preservation is a major determinant of initial graft function and survival. Graft viability is based on hypothermia, the organ being stored in a cold preservation solution.

Celsior® has been shown effective for cold preservation of heart and lung and, in laboratory studies, for liver, kidney and pancreas. The aim of the study is to evaluate the efficacy and safety of Celsior® in liver transplant preservation. Celsior® will be considered effective if the failure rate one year after transplantation is not significantly superior to 20% (rate observed in the European transplantation register between 1997 and 2001).

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Primary liver transplantation
* Whole organ transplantation
* Agreement for a 1 year follow-up
* Informed written consent

Exclusion Criteria:

* Liver disease secondary to clotting abnormalities
* Uncontrolled bacterial or viral disease at the time of transplantation
* Combined transplantations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-02; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Graft failure leading to patient death or retransplantation | 1 year

SECONDARY OUTCOMES:
Onset and severity of hemodynamic troubles at reperfusion | Reperfusion after transplantation
Onset of surgical complications | 1 year
Liver graft function during the fourteen first days | 14 days
Incidence, treatment and evolution of acute and chronic rejections histologically proven | 1 year
Onset of infections | 1 year
Onset, treatment and evolution of serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karim Boudjema, MD, PhD, Study Director — CHU Rennes; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (9):
- France (9):
  - Service de Chirurgie Digestive - Hôpital de la Côte de Nacre, Caen
  - Service de Chirurgie Digestive - Hôpital Henri Mondor, Créteil
  - Service de Chirurgie Viscérale et Transplantations - Hôpital Dupuytren, Limoges
  - Chirurgie générale et digestive - Hôpital de la Croix Rousse, Lyon
  - Service de Chirurgie Générale - Hôpital Edouard Herriot, Lyon
  - Service de Chirurgie Générale - Hôpital de la Conception, Marseille
  - Service de Chirurgie Générale et Digestive - Hôpital Cochin, Paris
  - Département de Chirurgie Viscérale - Hôpital Pontchaillou, Rennes
  - Service de Chirurgie Générale et Transplantation Multi-organe - Hôpital de la Hautepierre, Strasbourg

REFERENCES:
- [Background] Karam G, Compagnon P, Hourmant M, Despins P, Duveau D, Noury D, Boudjema K. A single solution for multiple organ procurement and preservation. Transpl Int. 2005 Jun;18(6):657-63. doi: 10.1111/j.1432-2277.2005.00083.x. PMID 15910289
- [Background] Adam R, Cailliez V, Majno P, Karam V, McMaster P, Caine RY, O'Grady J, Pichlmayr R, Neuhaus P, Otte JB, Hoeckerstedt K, Bismuth H. Normalised intrinsic mortality risk in liver transplantation: European Liver Transplant Registry study. Lancet. 2000 Aug 19;356(9230):621-7. doi: 10.1016/s0140-6736(00)02603-9. PMID 10968434